CLINICAL TRIAL: NCT06087835
Title: A Phase III, Randomised, Multicentre, Double-blind Study to Evaluate the Efficacy, Safety, and Tolerability of Zibotentan/Dapagliflozin Compared to Dapagliflozin Alone in Participants With Chronic Kidney Disease and High Proteinuria
Brief Title: Study to Investigate Efficacy, Safety, and Tolerability of Zibotentan/Dapagliflozin Compared to Dapagliflozin in Participants With Chronic Kidney Disease and High Proteinuria (ZENITH High Proteinuria)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4325C00010; 2023-504124-26 (Registry Identifier: EU CT number (CTIS))
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease With High Proteinuria
Keywords: Zibotentan; Nephrology; Dapagliflozin; Sodium-glucose co-transporter 2; sodium-glucose co-transporter 2 inhibitor; Kidney diseases; Endothelin antagonist; High Proteinuria
MeSH Terms: conditions — Kidney Diseases | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zibotentan/Dapagliflozin dose A or Zibotentan/Dapagliflozin dose B (Experimental): Drug dose (dose A or B) are determined based on eGFR values. Participants will receive daily oral dose of zibotentan/dapagliflozin in fixed dose combination.
  Interventions: Drug: Zibotentan/Dapagliflozin
- Dapagliflozin alone (Active Comparator): Participants will receive daily oral dose of dapagliflozin.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Zibotentan/Dapagliflozin — Participants will receive zibotentan/dapagliflozin in fixed-dose combination as per the arms they are randomized to
  Arms: Zibotentan/Dapagliflozin dose A or Zibotentan/Dapagliflozin dose B
Drug: Dapagliflozin — Participants will receive dapagliflozin as per the arms they are randomized to
  Arms: Dapagliflozin alone

SUMMARY:
This is a Phase III, randomised, multicentre, double-blinded study to evaluate efficacy, safety and tolerability of treatment with zibotentan/dapagliflozin and dapagliflozin alone in participants with chronic kidney disease (CKD) and high proteinuria

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age and of legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent.
2. Diagnosis of CKD, defined as eGFR ≥ 20 and < 90 mL/min/1.73 m2 and UACR > 700 mg/g (> 79 mg/mmol) or UPCR > 1000 mg/g (> 113 mg/mmoL).
3. All female participants must have a negative serum pregnancy test result at screening.
4. Female participants must be either

   * not of child-bearing potential or
   * women of child bearing potential (WOCBP) using at least one highly effective birth control method for at least 3 months prior to first dose of study intervention
5. Capable of giving signed informed consent
6. Provision of signed informed consent prior to any study specific procedure.
7. Provision of electronic informed consent prior to completion of the optional Study Participant Feedback Questionnaire (SPFQ).
8. Provision of signed and dated written Optional Genomics Initiative Research Information and Consent Form prior to collection of samples for optional genomics imitative research that supports the Genomic Initiative.
9. Receiving RAASi therapy (ACEi or ARB), and for the patient maximum tolerated labelled daily dose, that has been stable for at least 4 weeks.

Exclusion Criteria:

1. Participants with NYHA class III or class IV Congestive HF at the time of enrolment.
2. Participants hospitalised for HF during the last 6 month prior to screening.
3. Evidence of rales or jugular venous distention on physical examination.
4. Participants with type 1 diabetes mellitus.
5. History of any life-threatening ventricular dysrhythmia (continuous or paroxysmal).
6. Blood pressure above 160 mmHg systolic.
7. Blood pressure below 90 mmHg systolic.
8. Participants hospitalised for heart disease or cardiac procedures or for COVID-19 during the last 3 months prior to screening.
9. History of solid organ transplantation or bone marrow transplant.
10. History or ongoing allergy/hypersensitivity, as judged by the Investigator, to SGLT2i therapy (eg, dapagliflozin, canagliflozin, empagliflozin or other SGLT2 inhibitors) or Endothelin Receptor Antagonists (eg, ambrisentan, atrasentan, bosentan, or other).
11. Any condition with a life expectancy of less than 2 years based on investigator´s clinical judgment.
12. Malignancy within the past 5 years. Exceptions to this criterion include non-melanoma skin cancer and curatively treated cervical carcinoma in situ.
13. Significant liver disease as judged by the investigator or severe hepatic impairment with AST or ALT > 3 × ULN; or total bilirubin > 2 × ULN at time of screening. An isolated increase in bilirubin in participants with known Gilbert's syndrome is not a reason for exclusion.
14. Known blood-borne diseases.
15. Clinically significant, unstable, or uncontrolled medical condition as assessed by the Investigator.
16. Participants on renal replacement therapy or previous kidney transplant.
17. Known history of drug or alcohol abuse within 12 months of screening.
18. Participants on treatment with strong or moderate CYP3A4 inducer.
19. Participants on systemic immunosuppression therapy other than stable maintenance therapy defined as prednisone 10 mg/day (or equivalent) or less, aziothioprine 100 mg/day or less; MMF 1000 mg/day or less for at least 3 months prior to Visit 1. Inhaled, nasal or dermatological steroids are also allowed.
20. Participants treated or expecting to be treated with tolvaptan, any other ERAs, or budesonide (where used to treat IBD or IgAN).
21. Participation in another clinical study with a study intervention administered in the last 3 months.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1835 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Change in eGFR from baseline | At month 24
  To determine whether zibotentan and dapagliflozin in fixed dose combination is superior to dapagliflozin alone to slow decline in kidney function

SECONDARY OUTCOMES:
Change in Urine Albumin to Creatinine Ratio (UACR) from baseline to each participant's mean level | at Month 9
  To determine whether zibotentan and dapagliflozin in fixed dose combination is superior to dapagliflozin alone in reducing albuminuria
Time to the first occurrence of any of the components of the renal composite endpoint of 40% sustained decline in eGFR or ESKD or renal death | Through study completion, approximately 38 months
  To determine whether zibotentan and dapagliflozin in fixed dose combination is superior to dapagliflozin alone in reducing the incidence of the renal composite endpoint of 40% sustained decline in eGFR or ESKD or renal death
Change in Urine Protein to Creatinine Ratio (UPCR) from baseline to each participant's mean level | at Month 9
  To determine whether zibotentan and dapagliflozin in FDC is superior to dapagliflozin alone in reducing proteinuria in the biopsy-confirmed IgAN subgroup

CONTACTS AND LOCATIONS:
Locations (263):
- United States (58):
  - Research Site, Huntsville, Alabama
  - Research Site, Sun City West, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Huntington Park, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oxnard, California
  - Research Site, San Carlos, California
  - Research Site, San Dimas, California
  - Research Site, Tarzana, California
  - Research Site, Victorville, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jensen Beach, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Fayetteville, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Island Lake, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Bowling Green, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Silver Spring, Maryland
  - Research Site, Flint, Michigan
  - Research Site, Troy, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Albany, New York
  - Research Site, Middletown, New York
  - Research Site, Orchard Park, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Maumee, Ohio
  - Research Site, Pottstown, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Kingsport, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Mukilteo, Washington
  - Research Site, Spokane, Washington
- Argentina (3):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, Santa Fe
- Australia (5):
  - Research Site, Gosford
  - Research Site, Meadowbrook
  - Research Site, Perth
  - Research Site, Reservoir
  - Research Site, Southport
- Austria (2):
  - Research Site, Feldkirch
  - Research Site, Vienna
- Brazil (5):
  - Research Site, Belém
  - Research Site, Botucatu
  - Research Site, Joinville
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (5):
  - Research Site, Dobrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- China (28):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Deyang
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Linhai
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenzhen
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yantai
  - Research Site, Yibin
  - Research Site, Yinchuan
  - Research Site, Zhuzhou
  - Research Site, Zigong
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Roskilde
- France (8):
  - Research Site, La Tronche
  - Research Site, Mulhouse
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Rouen
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Tours
- Germany (7):
  - Research Site, Aachen
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, München
- India (5):
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Delhi
  - Research Site, Nadiād
  - Research Site, New Delhi
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (8):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Foggia
  - Research Site, Genoa
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Japan (33):
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Hashima-gun
  - Research Site, Kamakura-shi
  - Research Site, Kasuga-shi
  - Research Site, Kawaguchi-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kitakyusyu-shi
  - Research Site, Kofu
  - Research Site, Kurume-shi
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Matsumoto-shi
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Minokamo Shi
  - Research Site, Nishinomiya-Shi
  - Research Site, Nishinomiya-shi
  - Research Site, Okawa-shi
  - Research Site, Osaka
  - Research Site, Oyama-shi
  - Research Site, Sakushu
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Soka-shi
  - Research Site, Takamatsu
  - Research Site, Takasago-shi
  - Research Site, Tondabayashi-shi
  - Research Site, Toride-shi
  - Research Site, Urayasu
  - Research Site, Utsunomiya
- Malaysia (6):
  - Research Site, Alor Star
  - Research Site, Ipoh
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Seremban
  - Research Site, Seri Manjung
- Research Site, Mazatlán, Mexico
- Netherlands (3):
  - Research Site, Amersfoort
  - Research Site, Breda
  - Research Site, Dordrecht
- Norway (5):
  - Research Site, Bodø
  - Research Site, Lørenskog
  - Research Site, Oslo
  - Research Site, Stavanger
  - Research Site, Tromsø
- Poland (8):
  - Research Site, Chrzanów
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
- Slovakia (5):
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Púchov
  - Research Site, Rožňava
  - Research Site, Trebišov
- South Africa (7):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Chatsworth
  - Research Site, Durban
  - Research Site, Lenasia
  - Research Site, Midrand
  - Research Site, Parow
- South Korea (6):
  - Research Site, Ansan-si
  - Research Site, Busan
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chaingmai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Ratchathewi
- Turkey (Türkiye) (7):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Dinar
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- United Kingdom (5):
  - Research Site, Cardiff
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, York
- Vietnam (3):
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://vivli.org/

REFERENCES:
- [Derived] Smeijer JD, Wasehuus VS, Dhaun N, Gorriz JL, Soler MJ, Astrand M, Mercier AK, Greasley PJ, Ambery P, Heerspink HJL. Effects of Zibotentan Alone and in Combination with Dapagliflozin on Fluid Retention in Patients with CKD. J Am Soc Nephrol. 2024 Oct 1;35(10):1381-1390. doi: 10.1681/ASN.0000000000000436. Epub 2024 Jul 12. PMID 39352861